CLINICAL TRIAL: NCT01862549
Title: Adapting Dialectical Behavior Therapy for Children With Disruptive Mood Dysregulation Disorder: Pilot Randomized Clinical Trial
Brief Title: Adapting DBT for Children With DMDD: Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1205012350
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Disruptive Mood Dysregulation Disorder
MeSH Terms: interventions — Dialectical Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT for children (Experimental): Dialectical Behavior Therapy for children is a 32 session intervention (it consists of 2 pre-treatment sessions and 30 treatment sessions; treatment sessions are to be delivered in 32 weeks total) with once per week meetings, including 30 min. individual child therapy, 20 min. meeting with a caregiver and 40 min. of skills training with both.
  Interventions: Behavioral: Dialectical Behavior Therapy for children
- Treatment as Usual (Active Comparator): Children in active comparison conditions will receive Treatment as Usual (TAU) that primarily consists of 32 weekly sessions of supportive individual psychotherapy and adjunctive family interventions. Individual therapy included cognitive behavioral skills training (e.g., psychoeducation, cognitive modifications, thought blocking) and non-directive supportive therapy. Family therapy includes parenting skills training (e.g., limit setting, reinforcement techniques), structuring household environment, and safety planning.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy for children
  Arms: DBT for children
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
This study examines feasibility and preliminary efficacy of Dialectical Behavior Therapy adapted to children (DBT-C). DBT-C as compared to treatment-as-usual (TAU) is hypothesized to have lower drop-out rate, and higher treatment attendance and satisfaction. Further, DBT-C as compared to TAU will have significantly greater reduction in symptoms of Disruptive Mood Dysregulation disorder, including verbal and behavioral outbursts and angry/irritable mood.

DETAILED DESCRIPTION:
Specific Aims:

I: Conduct Pilot Randomized Clinical Trial to evaluate feasibility and efficacy of DBT for children with Disruptive Mood Dysregulation Disorder (DMDD) as compared with Treatment-As-Usual (TAU) (up to 30 children and caregivers in DBT-C and up to 30 children and caregivers in the treatment as usual comparison condition).

Specific Aim 1: Examine feasibility of DBT-C by evaluating the drop-out rates, number of session attended, and treatment satisfaction and any differences in these rates by groups, as well as therapist treatment adherence and competence.

Hypothesis 1: Attendance rate in DBT-C, as compared to TAU, will be at least 10% higher and drop-out rate will be at least 10% lower (primary feasibility endpoint). Further, DBT-C, as compared with TAU will have significantly higher treatment satisfaction rating by subjects (on the child and caregiver Therapy Satisfaction Questionnaires), and by therapists (on Therapist Satisfaction Scale), and higher patient compliance (on Psychosocial Treatment Compliance Scale). Therapist treatment adherence and competence as measured by DBT-C Treatment Integrity Scale, will not fall below 80%.

Specific Aim 2: Examine preliminary efficacy of DBT-C in reducing symptoms of Disruptive Mood Dysregulation Disorder.

Hypothesis 2: Children in DBT-C condition as compared to TAU will have significantly greater reduction in irritability, anger, aggression, temper outbursts, and mood instability (on Clinical Global Impression - Improvement scale [primary categorical outcome] Exploratory Aim 3: Examine efficacy of DBT-C in improving adaptive coping skills, emotional and behavioral regulation, social skills, and reducing aggressive behaviors, affective reactivity, non-suicidal self-harm behaviors, suicidal ideations, suicidal attempts, and non-suicidal self-harm urges.

Hypothesis 3: Children in DBT-C condition as compared to TAU will have significantly greater improvement in adaptive coping skills (on the Children's Coping Strategies Checklist), emotional and behavioral regulation (on the Emotion Regulation Checklist and Child Behavior Checklist - Dysregulation Syndrome) and social skills (on the Social Skills Rating Scale), and significantly greater reduction in aggressive behaviors (Measure of Aggression, Violence and Rage in Children), affective reactivity (on the Affective Reactivity Index and Mood Symptoms Questionnaire). ), and greater reduction in non-suicidal self-harm behaviors (in Columbia Suicide and Self-Injury Severity Rating Scale [C-SSIS] self-injurious behaviors), suicidal ideations (in the C-SSRS suicidal ideation classification category), suicidal attempts (in C-SSIS suicide attempts category), and non-suicidal self-harm urges (in C-SSIS self-injurious urges, no suicidal intent category).

Exploratory Aim 4: Examine efficacy of DBT-C in reducing the need for higher level services.

Hypothesis 4: Children in DBT-C condition as compared to TAU will have significantly fewer psychiatric hospitalization, emergency room visits, total number of days inpatient, and residential care placements (on the Services Assessment Form).

Exploratory Aim 5: Examine whether parent emotion regulation moderate the relationship between intervention and outcomes, while parent ability to effectively cope with children's negative emotions and children's coping skills and emotion regulation mediate outcomes.

Hypothesis 5: Parents' own emotion regulation (on the Difficulties in Emotion Regulation Scale) will moderate outcomes and parents' ability to effectively cope with children's negative emotions (on the Parental Response to Children's Negative Emotions), children coping skills (on the Children's Coping Strategies Checklist) and emotion regulation (on Emotion Regulation Checklist) will mediate outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 7 years 0 months to 12 years 11 months
2. Meet criteria for Disruptive Mood Dysregulation Disorder on DSM-IV
3. Stabilized on psychiatric medication (at least 6 weeks).
4. Able to be treated on the outpatient basis

Children with suicidal ideation, suicidal behavior and non-suicidal self-injury will be included (assessed using Columbia Suicide and Self-Injury Severity Rating Scale) unless other interventions are indicated (e.g., hospitalization, medication).

Exclusion Criteria:

1. Documented cognitive disability ( if records are not available will use < 85 IQ on Wechsler Intelligence Scale for Children-IV Information and Block Design subtests).
2. Current diagnosis of a psychotic disorder (on K-SADS-PL)
3. Pervasive Developmental Disorder (on K-SADS-PL)
4. Child in the English as Second Language program at school and/or caregivers have language difficulties as per self-report
5. Child is in state custody.
6. As consistent with DMDD diagnosis, child's co-morbid conditions better account for disruptive mood.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Attendance and drop-out rate measure | 32 weeks
Therapy Satisfaction Questionnaire | 32 weeks
Therapist Satisfaction Questionaire | 32 weeks
Psychosocial Treatment Compliance Scale | 32 weeks

SECONDARY OUTCOMES:
Clinical Global Impression Scale | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Mood Symptoms Questionnnaire | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Children Coping Strategies Checklist | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Emotion Regulation Checklist | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Child Behavior Checklist | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Social Skills Rating Scale | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Measure of Aggression, Violence and Rage in Children | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Affective Reactivity Index | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Columbia Suicide and Self-Injury Serevity Rating Scale | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Services Assessment Form | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Difficulties in Emotion Regulation Scale | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up
Parental Response to Children's Negative Emotions Scale | pre-treatment, 8, 16, 24, 32 weeks, 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francheska Perepletchikova, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States

REFERENCES:
- [Derived] Perepletchikova F, Nathanson D, Axelrod SR, Merrill C, Walker A, Grossman M, Rebeta J, Scahill L, Kaufman J, Flye B, Mauer E, Walkup J. Randomized Clinical Trial of Dialectical Behavior Therapy for Preadolescent Children With Disruptive Mood Dysregulation Disorder: Feasibility and Outcomes. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):832-840. doi: 10.1016/j.jaac.2017.07.789. Epub 2017 Aug 10. PMID 28942805
- See also: NCBI Link — http://www.ncbi.nlm.nih.gov/pubmed/21643467